CLINICAL TRIAL: NCT05775341
Title: Analysis of INtestinal Dysbiosis and TRanslocation of Bacteria in Patients Undergoing Abdominal Surgery
Brief Title: INtestinal Dysbiosis and TRanslocation of Bacteria in Patients Undergoing Surgery
Acronym: INTRA
Status: Active, not recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-01054
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — Mucosal swabs, intestinal mucosa and content, serum, mesenteric lymph node, subcutaneous biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — This is purely an observational study.

SUMMARY:
The goal of this observational study is to contribute to a better understanding of the perioperative kinetics of intestinal microbial composition and association with surgical site infections.

The main question this study aims to determine if:

* Patients undergoing surgery develop transient intestinal dysbiosis
* Such transient dysbiosis is associated with translocation to the systemic circulation and surgical site infection

Patients undergoing elective abdominal surgery will be included prospectively. Informed consent will be obtained. From patients the following information and samples will be collected:

* Perioperative: Baseline health data, nutrition data, measurement body composition, glucose monitoring
* Intraoperatively:

  * Mucosal swabs
  * Blood from central venous catheter and portal vein
  * Mesenteric lymph node
  * Intestinal specimen
  * Bile
  * Subcutaneous biopsy
* Postoperatively:

  * If a surgical site infection occurs samples from infected site

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing laparoscopic colorectal resection with anastomosis or patients undergoing duodeno-pancreatectomy.
* Elective surgery
* Informed consent
* Age > 18 years

Exclusion criteria:

* Emergency surgery
* Other surgery 30 days prior to surgery
* BMI <18 or >50kg/m2
* Planed simultaneous second procedure with involvement of the intestinal tract
* Cholestasis with cholangitis, hepatic disease (defined as cirrhosis Child B or C) or renal disease (acute or chronic renal failure defined as eGFR≤ 30ml/min)
* Severe active enteritis or colitis, malabsorption, enteric infections
* Pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective abdominal surgery
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of the intestinal microbiome between start and end of surgery | Day 0 (Day of Surgery)
  Score between PCA (principal components analysis) in the intestine between start (T1) and end (T2) of surgery.
  * Sampling: An intestinal specimen is dissected at start and end of elective pancreatic resections.
  * Processing: Samples are immediately processed for storage at -80° in glycerol.
  * Analysis: Quantification of total Biomass, DNA extraction, preparation of Bacterial DNA libraries, sequencing with Illumina system, downstream analysis, statistical analysis, principal components analysis (PCA) with all the samples is performed and the score is defined based on the distance between the two centers in PC1 and PC2 of T1 versus T2.

SECONDARY OUTCOMES:
Bacterial taxonomy in the intestine | Day 0 (Day of Surgery)
  Bacterial taxonomy in the intestine at start (T1) and end (T2) of surgery
Bacterial taxonomy MLN | Day 0 (Day of Surgery)
  Bacterial taxonomy MLN end (T2) of surgery
Bacterial taxonomy mucosal swabs | Day 0 (Day of Surgery)
  Bacterial taxonomy mucosal swabs at start (T1) and end (T2) of surgery
Bacterial taxonomy in the blood | Day 0 (Day of Surgery)
  Bacterial taxonomy in the blood at start (T1) and end (T2) of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Guido Beldi, Principal Investigator — Department of Visceral Surgery and Medicine, Bern University Hospital
Locations (1):
- Beldi Guido, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No